CLINICAL TRIAL: NCT00181207
Title: A Randomized, Sham-controlled, Double-blinded Pilot Study to Assess the Effects of High Frequency Chest Wall Oscillation (HFCWO) Therapy in Patients With Chronic Bronchitis
Brief Title: Airway Clearance for Prevention of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA_000202; 18-P-92858/3-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-02

CONDITIONS: COPD; Chronic Bronchitis; Emphysema
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Active (Experimental): Pneumatic Compression Device used twice daily for 20 minutes each time for 12 weeks
  Interventions: Device: pneumatic vest
- Sham (Placebo Comparator): Device looked and sounded like a pneumatic compression device, but was not inflating nor deflating.
  Interventions: Other: placebo pneumatic vest

INTERVENTIONS:
Device: pneumatic vest
  Arms: Active
Other: placebo pneumatic vest
  Arms: Sham

SUMMARY:
The purpose of this study is to show that one form of mechanical airway clearance techniques, High Frequency Chest Wall Oscillation (HFCWO)using a pneumatic vest, will diminish exacerbations of COPD which will improve respiratory health status.

DETAILED DESCRIPTION:
Approximately 60 to 70% of people with COPD have chronic cough and phlegm, the cardinal symptoms of chronic bronchitis or chronic mucus hypersecretion (CMH). Once thought to be a relatively benign condition, recent evidence shows that CMH in patients with established COPD is associated with greater decline in lung function, more frequent respiratory infections, more frequent exacerbations and increased mortality.Using mechanical airway clearance techniques (The Vest) will diminish exacerbations of COPD which will improve respiratory health status.

Comparison: Patients randomly assigned to the vest will have fewer exacerbations of COPD,better quality of life and less health care use compared to patients assigned to a sham vest.

ELIGIBILITY:
Inclusion Criteria:

* Physician Diagnosis of COPD,chronic bronchitis and/or emphysema
* Forced Expiratory Volume in 1 second (FEV1)/ Forced Vital Capacity (FVC) < or = 70%
* FEV1 < or = 65%
* Current or former smoker > or = 20 pack years
* History of 1 or more COPD exacerbations in past 6 months necessitation hospitalization, Emergency Department (ED) visit, antibiotic or steroid prescription

Exclusion Criteria:

* Other lung diseases
* Co-morbid illnesses such as cancer, liver disease, cardiomyopathy
* Recent chest wall or abdominal trauma or surgery that would preclude using the vest

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-05; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory B Diette, M.D.,M.H.S, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham: Placebo Comparator: Sham Device looked and sounded like a pneumatic compression device, but was not inflating nor deflating
- Active: Experimental: Active Pneumatic Compression Device used twice daily for 20 minutes each time for 12 weeks
Period: Overall Study
Arm/Group | Sham | Active
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham: received sham version of VEST
- Active: received functional version of VEST
- Total: Total of all reporting groups
Arm/Group | Sham | Active | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.0) | 62.5 (7.4) | 62.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 17 | 23 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is the Rate of Exacerbations as Defined Using the Winnipeg Criteria.
Description: count of exacerbations per group per 12 weeks. An exacerbation was defined based on three major symptoms: increasing dyspnea, increasing sputum purulence and increasing sputum volume. Exacerbations were counted if there were at least 2 of these 3 symptoms.
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: exacerbations per 12 weeks
Arm/Group | Sham | Active
Number analyzed (Participants) | 24 | 26
exacerbations per 12 weeks | 5.5 [3 to 8] | 4 [2 to 8]

2. Secondary Outcome: Quality of Life
Description: The SF-36 is used to measure health related quality of life. It assesses eight health concepts and provides physical and mental health summary scores. The summary scores range from 0 to 100, with 0 representing the worst and 100 the best quality of life.
Time Frame: Change from baseline to 12 weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sham | Active
Number analyzed (Participants) | 24 | 26
units on a scale | 5 [-5 to 10] | 0 [-12.5 to 5]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sham | Active
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No